CLINICAL TRIAL: NCT05047367
Title: The Relationship of Psychological Factors and Sleep Quality With the Severity of Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Emel Güler, Asst Prof, Cumhuriyet University
Other Study IDs: 2021-01/39
Record Dates: First submitted 2021-08-06; First posted 2021-09-17 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Carpal Tunnel Syndrome; Depressive Symptoms; Sleepiness; Anxiety; Sleep; Pain, Neuropathic
Keywords: CTS,Psychological factors,Sleep quality,Daytime Sleepiness
MeSH Terms: conditions — Carpal Tunnel Syndrome; Depression; Sleepiness; Anxiety Disorders; Neuralgia | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single-group studies: A total of 149 patients diagnosed with CTS, 126 female and 23 male, were included in the study
  Interventions: Behavioral: cross-sectional survey study

INTERVENTIONS:
Behavioral: cross-sectional survey study — Beck Depression Scale, Beck Anxiety Scale for psychological evaluation, Visual Analogue Scale and PainDETECT Questionnaire for pain, Pittsburgh Sleep Quality Scale and Epworth Sleepiness Scale for sleep quality
  Other Names: all patients were filled out forms for sleep quality and psychological evaluation

SUMMARY:
The most common entrapment neuropathy symptoms, the diagnosis of CTS, is determined by examination findings and by means of the results of electro-diagnostic test. With an increase in disease severity, trap neuropathy, whose symptoms are more pronounced at night, negatively affects the daily life of the person. Deterioration in sleep quality may cause depression and anxiety. Conflicting results have been found in the studies related to these findings. However, no study was found in which daytime sleepiness was evaluated in terms of CTS. The investigators aim in this study is to evaluate the relationship between CTS severity and depression, anxiety, sleep quality and daytime sleepiness.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common peripheral neuropathy with an incidence of 2.7-4%. CTS, resulting from compression of the median nerve in the wrist, clinically progresses with tingling, numbness matching the nerve trace, and motor deficit in the presence of progressive nerve damage. Accordingly, the incidence of neuropathic pain is increasing. In addition to these symptoms mentioned, electro-diagnostic tests are used for diagnostic purposes and to determine the severity of nerve compression, and as a result, there are different types of classification, but most commonly CTS is classified as mild, moderate and severe. This classification is of great importance for the regulation of the follow-up and treatment protocol and making the association of existing complaints with the disease. Studies have shown that approximately 80% of CTS patients wake up at night due to numbness in the hand, resulting in deterioration in sleep quality. Impairment of sleep quality may cause increased sympathetic nervous system activity and awakening of physical and psychological stressors. Deterioration in sleep quality may cause depression and anxiety. Conflicting results have been found in the studies related to these findings. However, no study was found in which daytime sleepiness was evaluated in terms of CTS. The investigators aim in this study is to evaluate the relationship between CTS severity and depression, anxiety, sleep quality and daytime sleepiness. This study;149 patients with a diagnosis of CTS were prospectively included in the study. Electro-diagnostic test results were used to determine the severity of the disease. In this context, Boston CTS rating scale was used to evaluate the functional and symptomatic effects, Pittsburgh sleep quality scale and Epworth sleepiness scale were used to evaluate sleep quality and daytime sleepiness, and pain DETECT questionnaire was used to evaluate pain type.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years diagnosed with CTS.
* Patients who were mentally able to respond to the assessment questionnaires were also included

Exclusion Criteria:

* Clinical diagnosis of cervical radiculopathy/plexopathy findings
* Pregnancy
* Diabetes mellitus
* thyroid diseases
* amyloidosis
* collagen tissue diseases
* Obstructive sleep apnea
* History of the upper extremity trauma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with CTS
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Severity of Carpal Tunnel Syndrome | study completion,an average of six months
  Electromyography evaluation of patients
The correlation between severity of Carpal Tunnel Syndrome and psychological evaluation | study completion,an average of six months
  Beck Depression Scale, Beck Anxiety Scale will be used for psychological evaluation. ≤9 points are classified as normal,10-16 points as mild depression,17-29 points as moderate depression, and 30-63 points as severe depression.Beck Anxiety Scale will be used in anxiety interrogation. ≤9 points are classified as normal, 10-18 points as mild anxiety, 19-29 points as moderate anxiety, and 30-63 points as severe anxiety.
The correlation between severity of Carpal Tunnel Syndrome and pain intensity | study completion,an average of six months
  Visual Analog Scale will be used for pain intensity.It is scored between 0-10. =: no pain 10: defined as the most severe pain
The correlation between severity of Carpal Tunnel Syndrome and neuropathic pain | study completion,an average of six months
  PainDETECT Questionnaire will be used for neuropathic pain evaluation.The questionnaire score ranges from 0-35 points, and a score of 19 and above indicates the presence of neuropathic pain.
The correlation between severity of Carpal Tunnel Syndrome and sleep quality | study completion,an average of six months
  Pittsburgh Sleep Quality Scale will be used for sleep quality. Those who score ˃5 have poor sleep quality, and those who score ≤5 have "good sleep quality"
The correlation between severity of Carpal Tunnel Syndrome and sleepiness | study completion,an average of six months
  Epworth Sleepiness Scale will be used for sleepiness. It is scored between 0-28. As the total score increases, sleepiness increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Guler, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
the importance of the data obtained in the study will be shared after

REFERENCES:
- [Result] Rubin G, Orbach H, Rinott M, Rozen N. Relationship between electrodiagnostic findings and sleep disturbance in carpal tunnel syndrome: A controlled objective and subjective study. J Int Med Res. 2020 Feb;48(2):300060519862673. doi: 10.1177/0300060519862673. Epub 2019 Jul 18. PMID 31319726